CLINICAL TRIAL: NCT03859973
Title: A Phase II Randomized, Double-blinded, Placebo-controlled Parallel Group Trial to Examine the Efficacy and Safety of BI 425809 Once Daily With Adjunctive Computerized Cognitive Training Over 12 Week Treatment Period in Patients With Schizophrenia
Brief Title: This Study Tests Whether BI 425809 Together With Brain Training Using a Computer Improves Mental Functioning in Patients With Schizophrenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1346-0038; 2018-002740-82 (EudraCT Number)
Record Dates: First submitted 2019-02-25; First posted 2019-03-01 (Actual); Results first posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-10

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — BI 425809

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BI 425809 10 mg + Computerized Cognitive Training (Experimental)
  Interventions: Drug: BI 425809
- Placebo + Computerized Cognitive Training (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BI 425809 — Tablet
  Other Names: iclepertin
  Arms: BI 425809 10 mg + Computerized Cognitive Training
Drug: Placebo — Tablet
  Arms: Placebo + Computerized Cognitive Training

SUMMARY:
This is a study in adults with schizophrenia. The study tests whether a medicine called BI 425809 together with brain training improves mental abilities.

Participants take study medication once a day for 12 weeks. At the start of the study, the participants are put into 2 groups. It is decided by chance who gets into which group. One group gets BI 425809 tablets every day. The other group gets placebo tablets every day. Placebo tablets look like the BI 425809 tablets, but contain no medicine. During the study, all participants do brain training using a computer.

The doctors regularly test mental abilities of the participants. The results of the mental ability tests are compared between the groups. The doctors also check the general health of the patients.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated written informed consent in accordance with ICH Harmonized Tripartite Guideline for Good Clinical Practice (ICH-GCP) and local legislation prior to admission to the trial.
* Male or female patients who are 18-50 years (inclusive) of age at time of consent.
* Established schizophrenia (as per DSM-5) with the following clinical features:

  * Outpatient, with no hospitalization for worsening of schizophrenia within 3 months prior to randomization
  * Psychiatrically stable without symptom exacerbation within 3 months prior to randomization
  * PANSS score ≤ 5 on positive items P1, P3-P7 and ≤ 4 on positive item P2 at Visit 1, and confirmed at Visit 2
* Patients must be on stable antipsychotic treatment; also, current antipsychotic medications and concomitant anticholinergics, antiepileptics, lithium and allowed antidepressants must meet the criteria below:

  * Patients must take 1 and may take up to 2 antipsychotics (typical and/or atypical), except for clozapine
  * Patients must be stable on current antipsychotics, anticholinergics, antiepileptics, lithium and allowed antidepressants for at least 3 months prior to randomization and be on current dose for at least 30 days prior to randomization o Patients on Long-Acting Injectable (LAI) antipsychotics should be on the same medication and dose for at least 3 months prior to randomization
* Women of childbearing potential (WOCBP)2 must be ready and able to use highly effective methods of birth control per Non-Clinical Safety Studies for the Conduct of Human Clinical Trials and Marketing Authorization for Pharmaceuticals (ICH M3 (R2)) that result in a low failure rate of less than 1% per year when used consistently and correctly. A list of contraception methods meeting these criteria is provided in Section 4.2.2.3. Such methods should be used throughout the trial, and for a period of at least 35 days after last trial drug intake, and the patient must agree to periodic pregnancy testing during participation in the trial.
* Patients must demonstrate their ability to properly use the CCT device and program, as well as be compliant with CCT run-in (defined as completing at least 2 hours per week for two weeks, totalling 4 hours CCT, during the screening period)3.
* Patients must be able to comply with all protocol procedures, in the investigator's opinion.
* Patients must have a study partner who will preferably be consistent throughout the study. It is recommended that the study partner should interact (in-person or telephone) with the subject at least 2 times a week.

Exclusion Criteria:

* Patients who have a categorical diagnosis of another current major psychiatric disorder on the Mini-International Neuropsychiatric Interview (M.I.N.I.).
* Diseases of the central nervous system (CNS) that may impact the assessment of the cognitive tests as per investigator's opinion. A movement disorder due to antipsychotic treatment not currently controlled with anti- EPS treatment or another movement disorder (e.g. Parkinson´s disease).
* Patients with a history of participating in any formal cognitive remediation program for 10 or more training sessions.
* Patients who were treated with any of the following medications within the last 6 months prior to randomization:

  * Bitopertin, BI 409306, encenicline or other investigational drug testing effects on cognition in schizophrenia
  * Clozapine (atypical antipsychotic medication)
  * Sarcosine, cycloserine, serine and glycine
  * Stimulants (e.g. methylphenidate, dextroamphetamine, modafinil)
  * Tricyclic antidepressants
* Patients receiving any other investigational drug (other than a potential cognitive enhancing drug) within 30 days or 6 half-lives (whichever is longer) prior to randomization. For investigational LAI antipsychotics, the last injection must be at least 3 months or two administration cycles (i.e. 6 months if administration is every 3 months) prior to randomization, whichever is longer.
* Patients who have participated in a clinical trial with repeated assessments (i.e. a single assessment is not exclusionary) with the MATRICS Consensus Cognitive Battery (MCCB) within the last 6 months prior to randomization.
* Patients who required a change in ongoing benzodiazepine or sleep medication dose or regimen within the last 30 days prior to randomization.
* Patients with known active infection with SARS-CoV-2 within the last 30 days prior to randomization.
* Other exclusion criteria apply

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-11-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (50):
- United States (28):
  - Atria Clinical Research, Little Rock, Arkansas
  - Woodland Research Northwest, Rogers, Arkansas
  - Encino Hospital Medical Center, Encino, California
  - Collaborative Neuroscience Network, LLC (CNS), Garden Grove, California
  - Synergy San Diego, Lemon Grove, California
  - Catalina Research Institute, LLC, Montclair, California
  - Pacific Research Partners, LLC, Oakland, California
  - NRC Research Institute, Orange, California
  - CNRI - Los Angeles, Pico Rivera, California
  - CNRI-San Diego, LLC, San Diego, California
  - Collaborative Neuroscience Network, LLC (CNS), Torrance, California
  - Meridien Research, Maitland, Florida
  - Premier Clinical Research Institute, Miami, Florida
  - University of Miami, Miami, Florida
  - Apalachee Center, Tallahassee, Florida
  - Jerome Golden Center for Behavioral Health, West Palm Beach, Florida
  - Synexus, Atlanta, Georgia
  - Uptown Research Institute, Chicago, Illinois
  - Lake Charles Clinical Trials LLC, Lake Charles, Louisiana
  - Cherry Health, Grand Rapids, Michigan
  - Center for Behavioral Medicine, Kansas City, Missouri
  - Synexus Clinical Research US, Inc., New York, New York
  - UNC Center for Excellence in Community Mental Health, North Carolina Psychiatric Research Center, Raleigh, North Carolina
  - Midwest Clinical Research, Dayton, Ohio
  - FutureSearch Trials of Dallas, LP, Dallas, Texas
  - Pillar Clinical Research, LLC, Richardson, Texas
  - Office of Dr. Aqeel Hashmi, MD, PA, Richmond, Texas
  - Northwest Clinical Research Center, Bellevue, Washington
- Australia (4):
  - Lyell McEwin Hospital, Elizabeth Vale, South Australia
  - Monash Medical Centre, Clayton, Victoria
  - St Vincent's Hospital Melbourne, Fitzroy, Victoria
  - Monash Alfred Psychiatry Research Centre, Melbourne, Victoria
- Canada (4):
  - University of Calgary, Calgary, Alberta
  - BC Mental Health and Addictions Research Institute (University of British Columbia), Vancouver, British Columbia
  - Centre for Addiction and Mental Health (CAMH), Toronto, Ontario
  - IUSMM Institut Universitaire en Sante Mentale de Montreal, Montreal, Quebec
- France (8):
  - CTR Esquirol, Caen
  - HOP Dijon-Bourgogne, Dijon
  - CAB Médical Psyché, Douai
  - HOP la Colombière, Montpellier
  - HOP Saint-Jacques, Nantes
  - HOP Pasteur, Nice
  - GHU Paris Psychiatrie et Neurosciences, Paris
  - HOP Nord, Saint-Priest-en-Jarez
- North Shore Hospital, Takapuna, Takpuna Auckland, New Zealand
- United Kingdom (5):
  - The Fritchie Centre, Cheltenham
  - Royal Edinburgh Hospital, Edinburgh
  - Queen Elizabeth University Hospital, Glasgow
  - Maudsley Hospital, London
  - Warneford Hospital, Oxford

IPD SHARING:
Plan to Share IPD: Yes
After the study is completed and the primary manuscript is accepted for publishing, researchers can use this following link https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement".
  Also, Researchers can use the following link https://www.mystudywindow.com/msw/datasharing to find information in order to request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
  The data shared are the raw clinical study data sets.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After all regulatory activities are completed in the US and EU for the product and indication, and after the primary manuscript has been accepted for publication.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'. For study data - 1. after the submission and approval of the research proposal (checks will be performed by both the independent review panel and the sponsor, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a 'Data Sharing Agreement'.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- [Derived] Harvey PD, McDonald S, Fu E, Reuteman-Fowler C. Efficacy and safety of iclepertin (BI 425809) with adjunctive computerized cognitive training in patients with schizophrenia. Schizophr Res Cogn. 2024 Dec 14;40:100340. doi: 10.1016/j.scog.2024.100340. eCollection 2025 Jun. PMID 39759424
- [Derived] Harvey PD, Bowie CR, McDonald S, Podhorna J. Evaluation of the Efficacy of BI 425809 Pharmacotherapy in Patients with Schizophrenia Receiving Computerized Cognitive Training: Methodology for a Double-blind, Randomized, Parallel-group Trial. Clin Drug Investig. 2020 Apr;40(4):377-385. doi: 10.1007/s40261-020-00893-8. PMID 32036587
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled in the trial once informed consent had been signed. Patients underwent computerised cognitive training (CCT) run-in for 2 weeks during the screening period. Patients compliant with the CCT run-in procedure and otherwise suitable after screening were randomised to the 12-week treatment period assigned at a ratio of 1:1 to 1 of 2 arms.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Groups:
- BI 425809 10 mg + Computerized Cognitive Training: Patients administered once daily (in the morning) two tablets of 5 milligram (mg) of BI 425809 (total BI 425809 dose= 10 mg) orally for 12 weeks. Concomitantly patients received non-pharmacological adjunctive computerized cognitive training (CCT).
- Placebo + Computerized Cognitive Training: Patients administered once daily (in the morning) two tablets of Placebo matching BI 425809 5 milligram (mg) orally for 12 weeks. Concomitantly patients received non-pharmacological adjunctive computerized cognitive training (CCT).
Period: Overall Study
Arm/Group | BI 425809 10 mg + Computerized Cognitive Training | Placebo + Computerized Cognitive Training
Started | 99 | 101
Completed (Completed trial medication) | 79 | 75
Not Completed | 20 | 26
Not completed — Other reason than listed | 3 | 2
Not completed — COVID-19 related, not due to AE | 3 | 4
Not completed — Withdrawal by Subject | 8 | 9
Not completed — Lost to Follow-up | 2 | 3
Not completed — Protocol Violation | 1 | 3
Not completed — Adverse Event | 3 | 5

BASELINE CHARACTERISTICS:
Population: Treated Set (TS) includes all patients in randomized set (RS) who were treated with at least 1 dose of the trial regimen (including both trial drug and computerized cognitive training (CCT)).
Groups:
- Total: Total of all reporting groups
Arm/Group | BI 425809 10 mg + Computerized Cognitive Training | Placebo + Computerized Cognitive Training | Total
Number analyzed (Participants) | 99 | 101 | 200
Age, Continuous [Mean (Standard Deviation); unit: Years] | 37.9 (8.1) | 38.5 (7.7) | 38.2 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 30 | 64
  Male | 65 | 71 | 136
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 16 | 28
  Not Hispanic or Latino | 87 | 85 | 172
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 4 | 5 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 44 | 40 | 84
  White | 47 | 51 | 98
  More than one race | 2 | 2 | 4
  Unknown or Not Reported | 2 | 0 | 2
Baseline MCCB neurocognitive composite T-score [Mean (Standard Deviation); unit: T-score] — Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) Consensus Cognitive Battery (MCCB) neurocognitive composite T-score assesses 6 cognitive domains, including speed of processing, attention vigilance, working memory, verbal learning, visual learning, reasoning and problem solving. MCCB neurocognitive T-scores in the general population have a mean of 50 and standard deviation of 10. A higher T-score indicates better cognition. Population: Treated Set (TS) includes all patients in randomized set (RS) who were treated with at least 1 dose of the trial regimen (including both trial drug and computerized cognitive training (CCT)). For one patient MCCB neurocognitive T-Score at baseline was not measured.
  T-score
    number analyzed (Participants) | 99 | 100 | 199
    (all) | 33.5 (12.0) | 34.0 (11.3) | 33.7 (11.6)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Neurocognitive Function as Measured by the Neurocognitive Composite Score of the Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) Consensus Cognitive Battery (MCCB) After 12 Weeks of Treatment
Description: MCCB neurocognitive composite T-score assesses 6 cognitive domains, including speed of processing, attention vigilance, working memory, verbal learning, visual learning, reasoning and problem solving. MCCB neurocognitive T-scores in the general population have a mean of 50 and standard deviation of 10. A higher T-score indicates better cognition. Change from baseline in MCCB neurocognitive composite T-score at Week 12 was modelled based on a restricted maximum likelihood (REML) based approach using a mixed model with repeated measurements (MMRM) which included the following fixed effects: categorical factor of planned treatment, visit (screening, baseline, week 6 and Week 12), planned treatment by visit interaction, continuous covariate of baseline value, baseline by visit interaction, categorical factor of age group, and continuous covariate of change from screening to baseline value. The Least Squares Mean (95 % Confidence Interval) at Week 12 is reported.
Time Frame: At screening (28 days prior to first drug drug administration), at baseline and at Weeks 6 and 12 after first drug administration.
Population: Full Analysis Set (FAS) includes all patients in treated set (TS) who had non-missing baseline and at least 1 non-missing post-baseline on-treatment measurement of the primary efficacy endpoint. The FAS was used for efficacy analyses. Patients were analysed as randomised.
Measure: Least Squares Mean (95% Confidence Interval); unit: T-score
Arm/Group | BI 425809 10 mg + Computerized Cognitive Training | Placebo + Computerized Cognitive Training
Number analyzed (Participants) | 88 | 86
T-score | 1.580 [0.370 to 2.790] | 2.466 [1.246 to 3.686]
Statistical Analysis 1: Comparison: BI 425809 10 mg + Computerized Cognitive Training vs Placebo + Computerized Cognitive Training; Restricted maximum likelihood (REML) based approach using a mixed model with repeated measurements (MMRM) which included the following fixed effects: categorical factor of planned treatment, visit (screening, baseline, week 6 and Week 12), planned treatment by visit interaction, continuous covariate of baseline value, baseline by visit interaction, categorical factor of age group, and continuous covariate of change from screening to baseline value; Test type: Other; p = 0.3101, Mixed Models Analysis; Mean Difference (Net) = -0.866, 95% CI 2-sided [-2.605 to 0.833] — Least Square Mean of (BI 425809 10 mg + Computerized Cognitive Training) - Least Square Mean of (Placebo + Computerized Cognitive Training)

2. Secondary Outcome: Change From Baseline in Cognitive Function as Measured by the Overall MCCB Composite T Score (Including Social Cognition) After 12 Weeks of Treatment
Description: MCCB cognitive score comprises 10 tests, which assess 7 cognitive domains, including speed of processing, attention vigilance, working memory, verbal learning, visual learning, reasoning and problem solving, and social cognition. MCCB cognitive T-scores in the general population have a mean of 50 and standard deviation of 10. A higher T-score indicates better cognition. Change from baseline in MCCB overall composite T-score was modelled using a restricted maximum likelihood (REML) based approach using a mixed model with repeated measurements (MMRM) which included the following fixed effects: categorical factor of planned treatment, visit (screening, baseline, week 6 and Week 12), planned treatment by visit interaction, continuous covariate of baseline value, baseline by visit interaction, categorical factor of age group, and continuous covariate of change from screening to baseline value. The Least Squares Mean (95 % Confidence Interval) at Week 12 is reported.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: T-score
Arm/Group | BI 425809 10 mg + Computerized Cognitive Training | Placebo + Computerized Cognitive Training
Number analyzed (Participants) | 88 | 86
T-score | 1.184 [-0.031 to 2.398] | 2.235 [1.011 to 3.459]
Statistical Analysis 1: Comparison: BI 425809 10 mg + Computerized Cognitive Training vs Placebo + Computerized Cognitive Training; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.2309, Mixed Models Analysis; Mean Difference (Net) = -1.051, 95% CI 2-sided [-2.778 to 0.676] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Change From Baseline in the Effect of Cognitive Deficit on Day-to-day Functioning as Measured by SCoRS Total Score After 12 Weeks of Treatment
Description: Schizophrenia Cognition Rating Scale (SCoRS) is a 20-item interview-based assessment of cognitive deficits and the degree to which they affect day-to-day functioning. Each item is rated on a 4-point scale. SCoRS total score is between 20 and 80 where higher score values represent greater degree of impairment in day-to-day functions due to cognitive deficits. The composite score was the average of non-missing responses. If five or more of the 20 items were missing, the composite score was missing for that participant at the visit.
  Change from baseline in SCoRS total score after 12 weeks of treatment was modelled using an Analysis of Covariance (ANCOVA) which included the following fixed effects: categorical factor of planned treatment, continuous covariate of baseline value, categorical factor of age group.
Time Frame: At baseline and at 12 weeks after first drug administration.
Population: Full Analysis Set (FAS) includes all patients in treated set (TS) who had non-missing baseline and at least 1 non-missing post-baseline on-treatment measurement of the primary efficacy endpoint. The FAS was used for efficacy analyses. Patients were analysed as randomised. Only patients with non-missing results at Week 12 are reported.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | BI 425809 10 mg + Computerized Cognitive Training | Placebo + Computerized Cognitive Training
Number analyzed (Participants) | 82 | 75
units on a scale | -2.495 [-3.724 to -1.266] | -3.072 [-4.358 to -1.787]
Statistical Analysis 1: Comparison: BI 425809 10 mg + Computerized Cognitive Training vs Placebo + Computerized Cognitive Training; Analysis of Covariance (ANCOVA) which included the following fixed effects: categorical factor of planned treatment, continuous covariate of baseline value, categorical factor of age group; Test type: Other; p = 0.5237, ANCOVA; Mean Difference (Net) = 0.577, 95% CI 2-sided [-1.207 to 2.362] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Change From Baseline in Positive and Negative Syndrome Scale (PANSS) Total Score After 12 Weeks of Treatment
Description: PANSS was used to evaluate broad psychopathology associated with schizophrenia disease state. The PANSS has 30 items. Each is rated from 1 to 7 points. The total factor score is the summation of the actual points for each item, leading the total score ranging from 30 to 210; a higher score indicates a worse disease condition.
  Change from baseline in PANNS total score after 12 weeks of treatment was modelled based on a restricted maximum likelihood (REML) based approach using a mixed model with repeated measurements (MMRM) which included the following fixed effects: categorical factor of planned treatment, visit (baseline, Week 6 and Week 12), planned treatment by visit interaction, continuous covariate of baseline value, baseline by visit interaction, categorical factor of age group. The Least Squares Mean (95 % Confidence Interval) at Week 12 is reported.
Time Frame: At baseline and at Weeks 6 and 12 after first drug administration.
Population: Full Analysis Set (FAS) includes all patients in treated set (TS) who had non-missing baseline and at least 1 non-missing post-baseline on-treatment measurement of the primary efficacy endpoint. The FAS was used for efficacy analyses. Patients were analysed as randomised. One patient in the arm "Placebo + Computerized Cognitive Training" was excluded from the statistical model, because the patient did not have post-baseline PANSS total score values.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | BI 425809 10 mg + Computerized Cognitive Training | Placebo + Computerized Cognitive Training
Number analyzed (Participants) | 88 | 85
units on a scale | -2.749 [-4.732 to -0.765] | -2.080 [-4.104 to -0.055]
Statistical Analysis 1: Comparison: BI 425809 10 mg + Computerized Cognitive Training vs Placebo + Computerized Cognitive Training; Restricted maximum likelihood (REML) based approach using a mixed model with repeated measurements (MMRM) which included the following fixed effects: categorical factor of planned treatment, visit (baseline, Week 6 and Week 12), planned treatment by visit interaction, continuous covariate of baseline value, baseline by visit interaction, categorical factor of age group; Test type: Other; p = 0.6420, Mixed Models Analysis; Mean Difference (Net) = -0.669, 95% CI 2-sided [-3.510 to 2.172] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Percentage of Patients With Any Adverse Event (AE) and With Serious Adverse Events (SAEs)
Description: Percentage of patients with any Adverse Event (AE) and with serious adverse events (SAEs) is reported.
  Percentages were rounded to one decimal place.
Time Frame: From first dose of study drug administration until four weeks after the last dose of study drug administration, up to 16 weeks.
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | BI 425809 10 mg + Computerized Cognitive Training | Placebo + Computerized Cognitive Training
Number analyzed (Participants) | 99 | 101
percentage of participants
  Any adverse event | 39.4 | 56.4
  Serious adverse events | 1.0 | 2.0

ADVERSE EVENTS:
Time Frame: From first dose of study drug administration until four weeks after the last dose of study drug administration, up to 16 weeks.
Description: Treated Set (TS) includes all patients in randomized set (RS) who were treated with at least 1 dose of the trial regimen (including both trial drug and computerized cognitive training (CCT)).
Arm/Group | BI 425809 10 mg + Computerized Cognitive Training | Placebo + Computerized Cognitive Training
All-Cause Mortality (participants affected / at risk) | 0/99 | 0/101
Serious Adverse Events (participants affected / at risk) | 1/99 | 2/101
Other Adverse Events (participants affected / at risk) | 9/99 | 16/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BI 425809 10 mg + Computerized Cognitive Training (N=99) | Placebo + Computerized Cognitive Training (N=101)
Colitis (Gastrointestinal disorders) | 1 | 0
COVID-19 (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Delirium (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BI 425809 10 mg + Computerized Cognitive Training (N=99) | Placebo + Computerized Cognitive Training (N=101)
Vomiting (Gastrointestinal disorders) | 3 | 6
Headache (Nervous system disorders) | 7 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2020-07-21): https://cdn.clinicaltrials.gov/large-docs/73/NCT03859973/Prot_000.pdf
  • Statistical Analysis Plan (2022-10-10): https://cdn.clinicaltrials.gov/large-docs/73/NCT03859973/SAP_001.pdf